CLINICAL TRIAL: NCT04182568
Title: Nab-paclitaxel Compared With Docetaxel Followed by Anthracyclines and Cyclophosphamide in the Neoadjuvant Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192081-F-1
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-paclitaxel (Experimental)
  Interventions: Drug: nab-paclitaxel followed by anthracycline and cyclophosphamide
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel followed by anthracycline and cyclophosphamide

INTERVENTIONS:
Drug: nab-paclitaxel followed by anthracycline and cyclophosphamide — nab-paclitaxel 260mg/m2 for every 2 weeks followed by anthracycline and cyclophosphamide
  Arms: nab-paclitaxel
Drug: Docetaxel followed by anthracycline and cyclophosphamide — Docetaxel 100 mg/m2 for for every 2 weeks followed by anthracycline and cyclophosphamide
  Arms: Docetaxel

SUMMARY:
This study is an open, multicenter, randomized controlled clinical trial for patients with newly diagnosed primary invasive breast cancer and clinical stage of T2 or above. The main purpose of this study is to evaluate the efficacy of dose-dense nab-paclitaxel compared with dose-dense docetaxel followed by anthracycline and cyclophosphamide in the treatment of HR positive and HER-2 negative breast cancer. The effectiveness and safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) age: 18-70 years old, female;

  2) patients with primary breast cancer, T2 or above, diagnosed by histopathology;

  3) HR was positive and HER-2 was negative by IHC;

  4) according to the RECIST 1.1 standard, there should be at least one measurable objective focus with tumor diameter > 2cm;

  5) ECoG physical fitness score 0-1;

  6) LVEF≥55%；

  7) bone marrow function: neutrophil ≥ 1.5 × 109 / L, platelet ≥ 100 × 109 / L, hemoglobin ≥ 90g / L;

  8) liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and alt ≤ 2.5 times the upper limit of normal value; total bilirubin ≤ 1.5 times the upper limit of normal value, or patients with Gilbert's syndrome ≤ 2.5 times the upper limit of normal value;

  9) patients have good compliance with the planned treatment, can understand the research process of this study and sign the written informed consent

Exclusion Criteria:

* 1) previously received cytotoxic chemotherapy, endocrine therapy, biological therapy or radiotherapy for any reason;

  2) patients with stage IV metastasis at the initial diagnosis;

  2) New York Heart Association (NYHA) rating of patients with heart disease above grade II (including grade II);

  3) patients with serious systemic infection or other serious diseases;

  4) patients who are known to be allergic or intolerant to chemotherapy drugs or their adjuvants;

  5) in the past 5 years, there have been other malignant tumors, except the cured carcinoma in situ of cervix and skin cancer without melanoma;

  6) pregnancy or lactation, as well as childbearing age patients who refuse to take appropriate contraceptive measures during the trial;

  7) participated in other experimental studies within 30 days before the administration of the first study drug;

  8) patients not suitable for the study were judged by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-08-21 (Estimated); Study Completion 2022-08-21 (Estimated)

PRIMARY OUTCOMES:
RCB | 2 years
  Residual tumor load

SECONDARY OUTCOMES:
pCR | 2 years
  Complete remission of Pathology

OTHER OUTCOMES:
DFS | 2 years
  Disease free survival
OS | 2 years
  Overall survival time

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China